CLINICAL TRIAL: NCT03551561
Title: Antisepsis Techniques in Orthopedic Surgical Procedures: a Comparative Study
Brief Title: Measures for the Prevention of Surgical Site Infection
Acronym: Orthopedics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Surgical Site Infection
Record Dates: First submitted 2018-04-08; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Infection
Keywords: Chlorhexidine; Infection; Orthopedics; Surgical rooms; Antisepsis; Surgical Procedures.
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CSAAC group (Active Comparator): The CSAAC group (chlorhexidine-based soap + ethyl alcohol + alcoholic chlorhexidine): skin preparation process with 4% chlorhexidine-based soap for a period of 5 minutes, followed by a sterile and soaked with 70% alcohol compress. After removing the chlorhexidine-based soap excess, antisepsis was performed with alcoholic chlorhexidine and surgical drapes and gowns. Cultures were performed in the mannitol and EMB (Eosin Methylene Blue) media after being collected at the pre-skin preparation, post-skin preparation process and end of the surgical procedure.
  Interventions: Drug: CSAAC; Drug: CSAC
- CSAC group (Active Comparator): The CSAC group (chlorhexidine-based soap + alcoholic chlorhexidine): skin preparation process with 4% chlorhexidine-based soap for a period of 5 minutes and the of a simple, dry and sterile compress to remove the excess. After removing the excess, antisepsis was performed with alcoholic chlorhexidine and surgical drapes and gowns. Cultures were performed in the mannitol and EMB media after being collected at the pre-skin preparation, post-skin preparation process and end of the surgical procedure.
  Interventions: Drug: CSAAC; Drug: CSAC

INTERVENTIONS:
Drug: CSAAC — Skin preparation with 4% chlorhexidine-based soap for a period of 5 minutes, followed by a sterile and soaked with 70% alcohol compress. After removing the chlorhexidine-based soap excess, antisepsis was performed with alcoholic chlorhexidine and surgical drapes and gowns.
  Other Names: chlorhexidine-based sopa+70% alcool+alcoholic chlorhexidine
Drug: CSAC — Skin preparation with 4% chlorhexidine-based soap for a period of 5 minutes and the of a simple, dry and sterile compress to remove the excess. After removing the excess, antisepsis was performed with alcoholic chlorhexidine and surgical drapes and gowns.
  Other Names: chlorhexidine-based sopa + alcoholic chlorhexidine

SUMMARY:
Among the causes associated with infection of hospitalized patients, surgical site infection is a complication that is potentially associated with any type of surgical procedure, it also represents an expressive burden in terms of morbidity and mortality, as well as additional costs for health care systems around the world. It is regarded that the efficiency of the pre, per, and postoperative skin preparation depends on both the adopted antiseptic and the application method, with Chlorhexidine currently being the most used drug in such preparation. However, the manner, timing, or timing of cutaneous antisepsis action is unclear. Objective: Comparing antisepsis techniques using chlorhexidine-based soap associated with ethyl alcohol and alcoholic chlorhexidine versus chlorhexidine-based soap associated with alcoholic chlorhexidine, in surgical orthopedic procedures.

DETAILED DESCRIPTION:
Among the causes associated with infection of hospitalized patients, surgical site infection is a complication that is potentially associated with any type of surgical procedure, it also represents an expressive burden in terms of morbidity and mortality, as well as additional costs for health care systems around the world. It is regarded that the efficiency of the pre, per, and postoperative skin preparation depends on both the adopted antiseptic and the application method, with Chlorhexidine currently being the most used drug in such preparation. However, the manner, timing, or timing of cutaneous antisepsis action is unclear. Objective: Comparing antisepsis techniques using chlorhexidine-based soap associated with ethyl alcohol and alcoholic chlorhexidine versus chlorhexidine-based soap associated with alcoholic chlorhexidine, in surgical orthopedic procedures. Methods: It is a primary, randomized, analytical and single-center clinical trial, consisting of 170 patients, which were distributed between 2 randomized groups, where Chlorhexidine-based Soap + Alcoholic Chlorhexidine were tested on the group CSAC and Chlorhexidine-based Soap + 70% Ethyl Alcohol + Alcoholic Chlorhexidine were tested on the group CSAAC. Cultures were performed in the Mannitol and EMB (Eosin Methylene Blue) media after being collected at the pre, post-skin preparation and end of the surgical procedure

ELIGIBILITY:
Inclusion Criteria:

* patients both males and females; older than 18 years old who will undergo orthopaedic surgical procedures;

Exclusion Criteria:

* patients who do not follow the medical guidelines; that are non-collaborative and / or do not sign the terms of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
Incidence of bacterial skin colonization | about 6 hours
  Skin culture

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio C Mendes, MD, Principal Investigator — Universidade do Vale do Sapucai
Locations (1):
- Universidade do Vale do Sapucai, Pouso Alegre, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bohl DD, Ondeck NT, Darrith B, Hannon CP, Fillingham YA, Della Valle CJ. Impact of Operative Time on Adverse Events Following Primary Total Joint Arthroplasty. J Arthroplasty. 2018 Jul;33(7):2256-2262.e4. doi: 10.1016/j.arth.2018.02.037. Epub 2018 Feb 17. PMID 29551302
- [Background] Capen DA, Calderone RR, Green A. Perioperative risk factors for wound infections after lower back fusions. Orthop Clin North Am. 1996 Jan;27(1):83-6. PMID 8539055
- [Background] Charles D, Heal CF, Delpachitra M, Wohlfahrt M, Kimber D, Sullivan J, Browning S, Saednia S, Hardy A, Banks J, Buttner P. Alcoholic versus aqueous chlorhexidine for skin antisepsis: the AVALANCHE trial. CMAJ. 2017 Aug 8;189(31):E1008-E1016. doi: 10.1503/cmaj.161460. PMID 28790056
- [Background] Cheng H, Chen BP, Soleas IM, Ferko NC, Cameron CG, Hinoul P. Prolonged Operative Duration Increases Risk of Surgical Site Infections: A Systematic Review. Surg Infect (Larchmt). 2017 Aug/Sep;18(6):722-735. doi: 10.1089/sur.2017.089. PMID 28832271
- [Background] Dicks KV, Baker AW, Durkin MJ, Anderson DJ, Moehring RW, Chen LF, Sexton DJ, Weber DJ, Lewis SS. Short Operative Duration and Surgical Site Infection Risk in Hip and Knee Arthroplasty Procedures. Infect Control Hosp Epidemiol. 2015 Dec;36(12):1431-6. doi: 10.1017/ice.2015.222. Epub 2015 Sep 22. PMID 26391277
- [Background] Drakos MC, Murphy CI. Bracing versus casting in ankle fractures. Phys Sportsmed. 2014 Nov;42(4):60-70. doi: 10.3810/psm.2014.11.2092. PMID 25419889
- [Background] Duchman KR, Pugely AJ, Martin CT, Gao Y, Bedard NA, Callaghan JJ. Operative Time Affects Short-Term Complications in Total Joint Arthroplasty. J Arthroplasty. 2017 Apr;32(4):1285-1291. doi: 10.1016/j.arth.2016.12.003. Epub 2016 Dec 14. PMID 28040399
- [Background] Ellenhorn JD, Smith DD, Schwarz RE, Kawachi MH, Wilson TG, McGonigle KF, Wagman LD, Paz IB. Paint-only is equivalent to scrub-and-paint in preoperative preparation of abdominal surgery sites. J Am Coll Surg. 2005 Nov;201(5):737-41. doi: 10.1016/j.jamcollsurg.2005.05.023. Epub 2005 Aug 31. PMID 16256917
- [Background] George J, Klika AK, Higuera CA. Use of Chlorhexidine Preparations in Total Joint Arthroplasty. J Bone Jt Infect. 2017 Jan 1;2(1):15-22. doi: 10.7150/jbji.16934. eCollection 2017. PMID 28529860
- [Background] Glassman SD, Dimar JR, Puno RM, Johnson JR. Salvage of instrumental lumbar fusions complicated by surgical wound infection. Spine (Phila Pa 1976). 1996 Sep 15;21(18):2163-9. doi: 10.1097/00007632-199609150-00021. PMID 8893444
- [Background] Hosseini P, Mundis GM Jr, Eastlack R, Nourian A, Pawelek J, Nguyen S, Akbarnia BA. Do Longer Surgical Procedures Result in Greater Contamination of Surgeons' Hands? Clin Orthop Relat Res. 2016 Jul;474(7):1707-13. doi: 10.1007/s11999-016-4832-1. Epub 2016 Apr 18. PMID 27090260
- [Background] Houang ET, Buckley R, Smith M, O'Riordan SM. Survival of Pseudomonas aeruginosa in plaster of Paris. J Hosp Infect. 1981 Sep;2(3):231-5. doi: 10.1016/0195-6701(81)90042-6. No abstract available. PMID 6174590
- [Background] Kamel C, McGahan L, Mierzwinski-Urban M, Embil J. Preoperative Skin Antiseptic Preparations and Application Techniques for Preventing Surgical Site Infections: A Systematic Review of the Clinical Evidence and Guidelines [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2011 Jun. Available from http://www.ncbi.nlm.nih.gov/books/NBK174549/ PMID 24354038
- [Background] Lee I, Agarwal RK, Lee BY, Fishman NO, Umscheid CA. Systematic review and cost analysis comparing use of chlorhexidine with use of iodine for preoperative skin antisepsis to prevent surgical site infection. Infect Control Hosp Epidemiol. 2010 Dec;31(12):1219-29. doi: 10.1086/657134. Epub 2010 Oct 22. PMID 20969449
- [Background] Levi AD, Dickman CA, Sonntag VK. Management of postoperative infections after spinal instrumentation. J Neurosurg. 1997 Jun;86(6):975-80. doi: 10.3171/jns.1997.86.6.0975. PMID 9171176
- [Background] Martinez J, Macias JH, Arreguin V, Alvarez JA, Macias AE, Mosqueda-Gomez JL. Isopropyl alcohol is as efficient as chlorhexidine to prevent contamination of blood cultures. Am J Infect Control. 2017 Apr 1;45(4):350-353. doi: 10.1016/j.ajic.2016.11.027. Epub 2017 Jan 12. PMID 28089672
- [Background] Mears SC, Dinah AF, Knight TA, Frassica FJ, Belkoff SM. Visibility of surgical site marking after preoperative skin preparation. Eplasty. 2008 Jul 16;8:e35. PMID 18709136
- [Background] Ovaska MT, Makinen TJ, Madanat R, Huotari K, Vahlberg T, Hirvensalo E, Lindahl J. Risk factors for deep surgical site infection following operative treatment of ankle fractures. J Bone Joint Surg Am. 2013 Feb 20;95(4):348-53. doi: 10.2106/JBJS.K.01672. PMID 23426769
- [Background] Peel TN, Cheng AC, Buising KL, Dowsey MM, Choong PF. Alcoholic Chlorhexidine or Alcoholic Iodine Skin Antisepsis (ACAISA): protocol for cluster randomised controlled trial of surgical skin preparation for the prevention of superficial wound complications in prosthetic hip and knee replacement surgery. BMJ Open. 2014 May 15;4(5):e005424. doi: 10.1136/bmjopen-2014-005424. PMID 24833699
- [Background] Prottey C, Pryce NG. Hand cleansing and skin condition. A comparison of conventional soap washing and the use of alcohol-impregnated paper cloths. Int J Cosmet Sci. 1987 Apr;9(2):53-8. doi: 10.1111/j.1467-2494.1987.tb00462.x. PMID 19456969
- [Background] Reichel M, Heisig P, Kohlmann T, Kampf G. Alcohols for skin antisepsis at clinically relevant skin sites. Antimicrob Agents Chemother. 2009 Nov;53(11):4778-82. doi: 10.1128/AAC.00582-09. Epub 2009 Sep 8. PMID 19738017
- [Background] Ridgeway S, Wilson J, Charlet A, Kafatos G, Pearson A, Coello R. Infection of the surgical site after arthroplasty of the hip. J Bone Joint Surg Br. 2005 Jun;87(6):844-50. doi: 10.1302/0301-620X.87B6.15121. PMID 15911671
- [Background] Roy-Camille R, Saillant G, Mazel C. Internal fixation of the lumbar spine with pedicle screw plating. Clin Orthop Relat Res. 1986 Feb;(203):7-17. PMID 3955999
- [Background] Saltzman MD, Nuber GW, Gryzlo SM, Marecek GS, Koh JL. Efficacy of surgical preparation solutions in shoulder surgery. J Bone Joint Surg Am. 2009 Aug;91(8):1949-53. doi: 10.2106/JBJS.H.00768. PMID 19651954
- [Background] Savage JW, Anderson PA. An update on modifiable factors to reduce the risk of surgical site infections. Spine J. 2013 Sep;13(9):1017-29. doi: 10.1016/j.spinee.2013.03.051. Epub 2013 May 24. PMID 23711958
- [Background] Schepers T, De Vries MR, Van Lieshout EM, Van der Elst M. The timing of ankle fracture surgery and the effect on infectious complications; a case series and systematic review of the literature. Int Orthop. 2013 Mar;37(3):489-94. doi: 10.1007/s00264-012-1753-9. Epub 2013 Jan 4. PMID 23288046
- [Background] Segal CG, Anderson JJ. Preoperative skin preparation of cardiac patients. AORN J. 2002 Nov;76(5):821-8. doi: 10.1016/s0001-2092(06)61035-1. PMID 12463081
- [Background] Veiga DF, Damasceno CAV, Veiga-Filho J, Figueiras RG, Vieira RB, Florenzano FH, Juliano Y, Ferreira LM. Povidone iodine versus chlorhexidine in skin antisepsis before elective plastic surgery procedures: a randomized controlled trial. Plast Reconstr Surg. 2008 Nov;122(5):170e-171e. doi: 10.1097/PRS.0b013e318186cd7f. No abstract available. PMID 18971711
- [Background] Vioreanu M, Dudeney S, Hurson B, Kelly E, O'Rourke K, Quinlan W. Early mobilization in a removable cast compared with immobilization in a cast after operative treatment of ankle fractures: a prospective randomized study. Foot Ankle Int. 2007 Jan;28(1):13-9. doi: 10.3113/FAI.2007.0003. PMID 17257532
- [Background] Weed S, Bastek JA, Sammel MD, Beshara M, Hoffman S, Srinivas SK. Comparing postcesarean infectious complication rates using two different skin preparations. Obstet Gynecol. 2011 May;117(5):1123-1129. doi: 10.1097/AOG.0b013e3182118e98. PMID 21508751

DOCUMENTS (1):
  • Informed Consent Form (2017-05-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT03551561/ICF_000.pdf